CLINICAL TRIAL: NCT07330154
Title: The Effectiveness of Nano Bio Fusion Gel (NBF) on Early Wound Healing at the Palate (Donor Site) After Soft Tissue Graft Surgery Compared to Placebo Gel: a Double Blinded Randomized Controlled Clinical Trial
Brief Title: The Effectiveness of Nano Bio Fusion Gingival Gel (NBF) on Wound Healing at the Palate (Donor Site) After Soft Tissue Graft Surgery Compared to Placebo Gel.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdullah University Hospital (Other)
Collaborators: Jordan University of Science and Technology (Other)
Responsible Party: Principal Investigator, Lana Bader, assistant professor, King Abdullah University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 440-2025; 2/185/2025 (Registry Identifier: Institutional Review Board at Jordan university of Science and Technology)
Record Dates: First submitted 2025-12-27; First posted 2026-01-09 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Wound Healing; Palatal Wound; Donor Site Complication; Inflammatory Cytokines
Keywords: NBF gel; wound healing; palatal donor site; soft tissue graft
MeSH Terms: interventions — Microscopy, Scanning Tunneling

STUDY DESIGN:
Intervention Model Description: The study will recriute patients require soft tissue graft surgery where the graft is harvested from the palate by free gingival graft or depithelized connective tissue graft, leaving an open wound in the palate (around 3×6 mm size) that is going to heal by secondary intesntion.
  They will be randomly assigned into 2 groups using computer generated randomization sequence:
  Group 1: placebo gel Group 2: NBF gel
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The gel will be provided in a small opaque tube. The clinician and the patient will be blinded to the type of gel used. Other doctor or dental assistant will be responsible for dispencing the gel to the patient according to the randomization sequence and the code sheet.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nano bio-fusion gingival gel (NBF) (Experimental): The gel should be applied 4 times daily for 4 weeks. After drying the surgical site in the palate with a sterile gauze, a pea size of the gel material is applied to the wound using cotton applicator. If there is a vertical relasing incision in the recipient site, the gel will be applied using the same technique.
  Interventions: Drug: Application of NBF gel after soft tissue graft surgery
- placebo gel (Placebo Comparator): The gel should be applied 4 times daily for 4 weeks. After drying the surgical site in the palate with a sterile gauze, a pea size of the gel material is applied to the wound using cotton applicator. If there is a vertical relasing incision in the recipient site, the gel will be applied using the same technique.
  Interventions: Other: Application of placebo gel after soft tissue graft surgery

INTERVENTIONS:
Drug: Application of NBF gel after soft tissue graft surgery — After the surgery, patients will be instructed to apply the NBF gel to the donor site on the palate for four times daily for 4 weeks. If there is a vertical releasing incision in the recipient site, the gel will be applied along that incision too. The first application will be performed immediately after surgery by the investigator using a sterile cotton applicator.
  Other Names: phenotype modification; recession coverage; free gingival graft; connective tissue graft; coronal position flap; subepithelial connective tissue graft; tunnelling; lateral position flap
  Arms: Nano bio-fusion gingival gel (NBF)
Other: Application of placebo gel after soft tissue graft surgery — After the surgery, patients will be instructed to apply the placebo gel to the donor site on the palate for four times daily for 4 weeks. If there is a vertical releasing incision in the recipient site, the gel will be applied along that incision too. The first application will be performed immediately after surgery by the investigator using a sterile cotton applicator.
  Other Names: phenotype modification; recession coverage; free gingival graft; connective tissue graft; coronal position flap; subepithelial connective tissue graft; tunnelling; lateral position flap
  Arms: placebo gel

SUMMARY:
The goal of this clinical trial is to assess the effect of Nano-biofusion gingival gel (NBF) on wound healing at the palatal donor site following soft tissue graft surgery and compare it to placebo gel. The main questions it aims to answer are:

* Does NBF gel enhance wound healing after graft harvesting from the palate?
* Does NBF gel reduce the number of inflammatory mediators after surgery?
* Does NBF gel reduce pain and discomfort at the palatal donor site? Researchers will compare NBF gel to a placebo (a look-alike gel that does not contain the active ingredients) to see if NBF gel enhances wound healing.

Study steps include:

* Participants will apply the assigned gel on the surgical wound 4 times a day for 4 weeks.
* Clinical photographs and measurements will be obtained on days (0, 1, 2, 4, 7, 15, 21, 30).
* Wound fluid samples will be collected on days (0, 1, 2, 4, 7).
* Participants will be asked about the level of pain and analgesic consumption on each follow-up visit.

DETAILED DESCRIPTION:
A sample size of 36 subjects, with treated 18 sites in each group should be sufficient to detect a mean difference of 1 mm of the wound area between groups. Efforts will be made to balance the number of men and women in each group (if possible).

The participants will be recruited from patients coming to dental teaching clinics at Jordan University of Science and Technology. The patients will be randomly assigned into 2 groups using computer generated randomization sequence:

Group 1: placebo gel Group 2: NBF gel

The study's purpose and procedures will be clearly communicated to all patient. Prior to examination and treatment, each participant must sign a consent form.

Patients who require a soft tissue surgery to cover gingival recession around teeth, to modify the phenotype where there is a thin gingival tissue, or to increase the width and thickness of soft tissue will be included in the study. The soft tissue graft should be obtained from the palatal donor site by free gingival graft or depithelized connective tissue graft, leaving an open wound in the palate (around 3×6 mm size) that is going to heal by secondary intesntion.

After the procedure, patients will be instructed to use the gel 4 times a day for 4 weeks by applying it to the wound and massaging the area. It will be provided in a small opaque tube. One tube should be used each day. The clinician and the patient will be blinded to the type of gel used. Another doctor or dental assistant will be responsible for dispencing the gel to the patient according to the randomization sequence and the code sheet.

Oral hygiene measures will be prohibited for the first 2 weeks in the surgical area only to not disturb the wound healing. Patients should follow their oral hygiene routine for the rest of the teeth. They will be instructed to use 0.2% chlorhexidine mouth wash twice a day for 2 weeks after surgery.

The study will last for one month for each patient. Each patient will be assessed immediately before and after the surgery and on days (0, 1, 2, 4, 7, 15, 21, 30). Clinical photographs will be taken at each time point.

Wound fluid samples (WF) will be collected at the incision area immediately after surgery and wound closure (day 0) and on days (1, 2, 4, 7). Main inflammotry mediators will be assessed.

Study steps:

• T0(intervention): Pt will sign the consent form. Sof tissue graft surgery will be performed and the graft will be obtained from the palate. The surgery is not performed by one periodontist, but the assessment and measurements are done by the same blinded examiner.

• T1 (24 hours after the surgery), T2 (2 days after the surgery), T3 (4 days after the surgery), T4 (7 days after the surgery), T5 (15 days after the surgery), T6 (21 days after the surgery), T7 (30 days after the surgery): The wound will be measured to record all the primary and secondary outcomes. The exception is made for the collection of wound fluid samples on days 15, 21 and 30. As the wound will be probably closed by then, samples will not be collected, unless there is delayed wound healing and the fluid can be drawn from the wound.

Clinical photos will be taken before surgery and anesthesia, immediately after surgery and the rest of time points.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with gingival recession that is indicated for root coverage or need for phenotype modification.
2. 18 years or older.
3. absence of systemic disease
4. Non-smoker
5. No use of antibiotics, corticosteroids, anti-inflammatory medication or hormones in the past 3 months

Exclusion Criteria:

1. Pregnant or lactating woman.
2. patients with immune or systemic diseases.
3. Patients with an allergy to any ingredient in the gel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-10-29 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Wound area | On each follow up visit: T1 (24 hours after the surgery), T2 (2 days after the surgery), T3 (4 days after the surgery), T4 (7 days after the surgery), T5 (15 days after the surgery), T6 (21 days after the surgery), T7 (30 days after the surgery)
  The wound area of the palatal donor site will have a rectangular shape, and it will be measured in mm according to the following equation:
  Area = length × width UNC15 periodontal probe will be used to do the measurements at the greatest dimension horizontally and vertically. The site will be left to heal by secondary intension.

SECONDARY OUTCOMES:
Early wound healing index (EWHI) | On each follow up visit: T1 (24 hours after the surgery), T2 (2 days after the surgery), T3 (4 days after the surgery), T4 (7 days after the surgery), T5 (15 days after the surgery), T6 (21 days after the surgery), T7 (30 days after the surgery)
  the amount of fibrin at the wound margin will be assessed using early wound healing index (EWHI). The index was used to assess healing after papilla preservation flap. It will be modified to use at the vertical releasing incision of the recipient site according to the following criteria:
  1. complete flap closure-no fibrin line at the incision line
  2. complete flap closure-fine fibrin line at the incision line
  3. complete flap closure-fibrin clot at the incision line
  4. incomplete flap closure-partial tissue necrosis at the incision line
  5. incomplete flap closure-complete tissue necrosis at the at the incision line
Present or abscent (Yes/no): | On each follow up visit: T1 (24 hours after the surgery), T2 (2 days after the surgery), T3 (4 days after the surgery), T4 (7 days after the surgery), T5 (15 days after the surgery), T6 (21 days after the surgery), T7 (30 days after the surgery)
  1. Pus discharge
  2. Bleeding on palpation
  3. Tenderness on palpation
  4. Presence of granulation tissue
  5. Scar (yes/no……if yes, wider or lesser than 2 mm, contour: regular or irregular)
Erythema, redness + edema, swelling | On each follow up visit: T1 (24 hours after the surgery), T2 (2 days after the surgery), T3 (4 days after the surgery), T4 (7 days after the surgery), T5 (15 days after the surgery), T6 (21 days after the surgery), T7 (30 days after the surgery)
  mild <50% of the wound area, moderate 50%, severe >50%.
Epithelization and exposure of CT | On each follow up visit: T1 (24 hours after the surgery), T2 (2 days after the surgery), T3 (4 days after the surgery), T4 (7 days after the surgery), T5 (15 days after the surgery), T6 (21 days after the surgery), T7 (30 days after the surgery)
  partial or complete epithelization
Incision margins | On each follow up visit: T1 (24 hours after the surgery), T2 (2 days after the surgery), T3 (4 days after the surgery), T4 (7 days after the surgery), T5 (15 days after the surgery), T6 (21 days after the surgery), T7 (30 days after the surgery)
  measured for the vertical incsion on the recipient site if present. It will be recorded as: merged, in contact or in distance.
Patient reported outcome measure (PROM) | On each follow up visit: T1 (24 hours after the surgery), T2 (2 days after the surgery), T3 (4 days after the surgery), T4 (7 days after the surgery), T5 (15 days after the surgery), T6 (21 days after the surgery), T7 (30 days after the surgery)
  Pain intensity: will be recorded on a visual analogue scale from 1-10. The higher the number the more the pain.
  * Duration: min, hour, whole day
  * Nature: continuous or intermittent - Consumption of Analgesics: Patients will be instructed to use 2 tabs of paracetamol 500 mg in case they feel pain. They should not use any other type of analgesics as it might affect the healing and inflammation. They will be requested to record the number of tablets and the times they were taken
cytokine measurement using ELISA test | Immediately after surgery and wound closure (day 0) and on days (1, 2, 4, 7). They will not be collected at days 15, 21, and 30 as the wound should be closed by then, unless there is delayed wound healing and the fluid can be collected from the wound.
  Wound fluid samples (WF) will be collected from the palatal donor site and at the vertical incision using sterile paper points. Levels of cytokines (IL-1β, TNF-α, IL-6, IL-10) will be determined with Enzyme-Linked immunosorbent Assay test (ELISA) following the manufacturer's instructions.

CONTACTS AND LOCATIONS:
Overall Officials: Lana Bader, DClinDent Perio, Study Director — Jordan University of Science and Technology; Rand Aldurra, MClinDent Perio, Principal Investigator — Jordan University of Science and Technology
Locations (1):
- Jordan University of Science and Technology, Faculty of Dentistry, Irbid, Irbid Governorate, Jordan

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data for wound size, early wound healing index, and patient-reported outcomes will be shared. Data will be stripped of all identifiers to protect participants privacy.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD and supporting documents will be available after publication of the main study results, for a period of one year.
Access Criteria: Access will be granted to qualified researchers who request the data via email to the principal investigator. Researchers must sign a data use agreement ensuring ethical use, confidentiality, and prohibition of attempts to identify participants.